CLINICAL TRIAL: NCT00239681
Title: A Randomized, Double-Blind, Placebo Controlled, Multicenter, Phase 3 Study of Rosuvastatin (CRESTOR®) 20 mg in the Prevention of Cardiovascular Events Among Subjects With Low Levels of Low Density Lipoprotein(LDL) Cholesterol & Elevated Levels of C-Reactive Protein
Brief Title: JUPITER - Crestor 20mg Versus Placebo in Prevention of Cardiovascular (CV) Events
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See detailed description for reason.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D3560L00030; Jupiter; 4522US/0011
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-02

CONDITIONS: Elevated High-sensitivity C-Reactive Protein (hsCRP)
Keywords: Primary prevention; Cardiovascular disease; Statin therapy; C-reactive protein
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Experimental): Rosuvastatin 20 mg once daily
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Oral
  Other Names: Crestor
  Arms: Rosuvastatin
Other: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of long-term therapy with rosuvastatin compared with a placebo, and to evaluate whether treatment with rosuvastatin might be effective in reducing the risk of major cardiovascular events.

DETAILED DESCRIPTION:
AstraZeneca announced it has decided to stop the CRESTOR JUPITER clinical study early based on a recommendation from an Independent Data Monitoring Board and the JUPITER Steering Committee, which met on March 29, 2008. The study will be stopped early because there is unequivocal evidence of a reduction in cardiovascular morbidity and mortality amongst patients who received CRESTOR when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men 50 years or older, women 60 years or older
* Low to normal levels of low density lipoprotein (LDL) cholesterol (< 130mg/dL)
* Elevated levels of C-Reactive Protein (CRP) > 2.0 mg/L

Exclusion Criteria:

* History of cardiovascular or cerebrovascular events
* Active liver disease
* Diabetes mellitus
* Uncontrolled hypertension or hypothyroidism
* History of certain malignancies
* Chronic inflammatory conditions
* History of alcohol or drug abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17802 (Actual)
Dates: Start 2003-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hsia, MD, Study Director — AstraZeneca; Paul Ridker, MD, Study Chair — Brigham and Women's Hospital
Locations (856):
- United States (431):
  - Research Site, Birmingham, Alabama
  - Research Site, Calera, Alabama
  - Research Site, Columbiana, Alabama
  - Research Site, Decatur, Alabama
  - Research Site, Graysville, Alabama
  - Research Site, Haleyville, Alabama
  - Research Site, Hartselle, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Muscle Shoals, Alabama
  - Research Site, South Birmingham, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Pine Bluff, Arkansas
  - Research Site, Alhambra, California
  - Research Site, Azusa, California
  - Research Site, Berkeley, California
  - Research Site, Beverly Hills, California
  - Research Site, Burlingame, California
  - Research Site, Carmichael, California
  - Research Site, Concord, California
  - Research Site, Culver City, California
  - Research Site, Daly City, California
  - Research Site, Folsom, California
  - Research Site, Foothill Ranch, California
  - Research Site, Fountain Valley, California
  - Research Site, Fresno, California
  - Research Site, Garden Grove, California
  - Research Site, Inglewood, California
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, La Mesa, California
  - Research Site, Languna Niguel, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Los Gatos, California
  - Research Site, Mission Hills, California
  - Research Site, Mission Viejo, California
  - Research Site, Modesto, California
  - Research Site, Newport Beach, California
  - Research Site, Norwalk, California
  - Research Site, Orange, California
  - Research Site, Orangevale, California
  - Research Site, Palm Desert, California
  - Research Site, Pasadena, California
  - Research Site, Pismo Beach, California
  - Research Site, Pomona, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, San Ramon, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, Upland, California
  - Research Site, Ventura, California
  - Research Site, Vista, California
  - Research Site, Walnut Creek, California
  - Research Site, Westlake Village, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Highlands Ranch, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Loveland, Colorado
  - Research Site, Avon, Connecticut
  - Research Site, Bristol, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Trumbull, Connecticut
  - Research Site, West Hartford, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Wlimington, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Apopka, Florida
  - Research Site, Beverly Hills, Florida
  - Research Site, Cape Coral, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Cooper City, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Davie, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Largo, Florida
  - Research Site, Margate, Florida
  - Research Site, Miami, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Sebastian, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Brunswick, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Conyers, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Fayetteville, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Aurora, Illinois
  - Research Site, Champaign, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Lake Road, Illinois
  - Research Site, Melrose Park, Illinois
  - Research Site, Morton, Illinois
  - Research Site, O'Fallon, Illinois
  - Research Site, Orland Park, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Sterling, Illinois
  - Research Site, Vernon Hills, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Granger, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Jeffersonville, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Newburgh, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Dubuque, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Leavenworth, Kansas
  - Research Site, Olathe, Kansas
  - Research Site, Overland Park, Kansas
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Evansville, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Houma, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Research Site, Marrero, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Portland, Maine
  - Research Site, Sanford, Maine
  - Research Site, South Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Charlotte Hall, Maryland
  - Research Site, Glen Burnie, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Prince Frederick, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ayer, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, East Bridgewater, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Natick, Massachusetts
  - Research Site, Newton, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, West Yarmouth, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Berkley, Michigan
  - Research Site, Dearborn, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Livonia, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Portage, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Warren, Michigan
  - Research Site, Chaska, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Gulfport, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Olive Branch, Mississippi
  - Research Site, Picayune, Mississippi
  - Research Site, Port Gibson, Mississippi
  - Research Site, Chesterfield, Missouri
  - Research Site, Excelsior Springs, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Manchester, Missouri
  - Research Site, Mexico, Missouri
  - Research Site, Rolla, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, Shawnee Mission, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Washington, Missouri
  - Research Site, Wentzville, Missouri
  - Research Site, Anaconda, Montana
  - Research Site, Butte, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Missoula, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Nashua, New Hampshire
  - Research Site, Bloomfield, New Jersey
  - Research Site, Brick, New Jersey
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Elizabeth, New Jersey
  - Research Site, Englewood Cliffs, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Northbrunswick, New Jersey
  - Research Site, Passaic, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Trenton, New Jersey
  - Research Site, West Caldwell, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Los Alamos, New Mexico
  - Research Site, Rio Rancho, New Mexico
  - Research Site, Albany, New York
  - Research Site, Binghamton, New York
  - Research Site, Bowmansville, New York
  - Research Site, Bronxville, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Camillus, New York
  - Research Site, East Islip, New York
  - Research Site, East Syracuse, New York
  - Research Site, Fayetteville, New York
  - Research Site, Lake Success, New York
  - Research Site, Mamaroneck, New York
  - Research Site, Mount Vernon, New York
  - Research Site, New Hartford, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Niagara Falls, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Riverhead, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Tonawanda, New York
  - Research Site, Williamsville, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Burlington, North Carolina
  - Research Site, Cary, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Lenoir, North Carolina
  - Research Site, Lexington, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Athens, Ohio
  - Research Site, Bellbrook, Ohio
  - Research Site, Canal Fulton, Ohio
  - Research Site, Centerville, Ohio
  - Research Site, Chesterland, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Wadsworth, Ohio
  - Research Site, Warren, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Guthrie, Oklahoma
  - Research Site, Muskogee, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Yukon, Oklahoma
  - Research Site, Corvallis, Oregon
  - Research Site, Dallas, Oregon
  - Research Site, Eugene, Oregon
  - Research Site, Lake Oswego, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Milwaukie, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Springfield, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Beaver, Pennsylvania
  - Research Site, Bloomsburg, Pennsylvania
  - Research Site, Broomall, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Connellsville, Pennsylvania
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Fleetwood, Pennsylvania
  - Research Site, Harleysville, Pennsylvania
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, King of Prussia, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Lansdowne, Pennsylvania
  - Research Site, Lewisburg, Pennsylvania
  - Research Site, Lewistown, Pennsylvania
  - Research Site, Lock Haven, Pennsylvania
  - Research Site, McMurray, Pennsylvania
  - Research Site, Melrose Park, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Plymouth Meeting, Pennsylvania
  - Research Site, Reading, Pennsylvania
  - Research Site, Scotland, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Souderton, Pennsylvania
  - Research Site, Springfield, Pennsylvania
  - Research Site, State College, Pennsylvania
  - Research Site, Stoneboro, Pennsylvania
  - Research Site, Tipton, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Wallingford, Pennsylvania
  - Research Site, Warminster, Pennsylvania
  - Research Site, West Grove, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Cranston, Rhode Island
  - Research Site, Johnston, Rhode Island
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Providence, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Hampton, South Carolina
  - Research Site, Moncks Corner, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Clarksville, Tennessee
  - Research Site, Fayetteville, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Jefferson City, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Morristown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Colleyville, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Friendswood, Texas
  - Research Site, Grapevine, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Lake Jackson, Texas
  - Research Site, Lubbock, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Pharr, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Seguin, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Tyler, Texas
  - Research Site, Bountiful, Utah
  - Research Site, Nephi, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont
  - Research Site, Alexandria, Virginia
  - Research Site, Arlington, Virginia
  - Research Site, Burke, Virginia
  - Research Site, Charlottesville, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Hayes, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Quinton, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Springfield, Virginia
  - Research Site, Stuart, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Weber City, Virginia
  - Research Site, Yorktown, Virginia
  - Research Site, Burien, Washington
  - Research Site, Everett, Washington
  - Research Site, Gig Harbor, Washington
  - Research Site, Olympia, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Lewisburg, West Virginia
  - Research Site, Beloit, Wisconsin
  - Research Site, Green Bay, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Menomonee Falls, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (10):
  - Research Site, Capital Federal, Buenos Aires
  - Research Site, Pilar, Buenos Aires
  - Research Site, Quilmes, Buenos Aires - Argentina
  - Research Site, Ramos Mejía, Buenos Aires Argentina
  - Research Site, San Isidro, Buenos Aires- Argentina
  - Research Site, Córdoba, Cordoba - Argentina
  - Research Site, Salta, Salta Province
  - Research Site, Rosario, Santa Fe- Argentina
  - Research Site, San Miguel de Tucumán, Tucuman / Argentina
  - Research Site, San Miguel de Tucumán, Tucuman-argentina
- Belgium (74):
  - Research Site, Alsemberg, Belgium
  - Research Site, Anthée, Belgium
  - Research Site, Auvelais, Belgium
  - Research Site, Baisy-Thy, Belgium
  - Research Site, Bertrix, Belgium
  - Research Site, Betekom, Belgium
  - Research Site, Boechout, Belgium
  - Research Site, Braine-l'Alleud, Belgium
  - Research Site, Burdinne, Belgium
  - Research Site, Cerexhe-Heuseux, Belgium
  - Research Site, Champion, Belgium
  - Research Site, Chênée, Belgium
  - Research Site, Comines, Belgium
  - Research Site, Deurne (antwerpen), Belgium
  - Research Site, Dour, Belgium
  - Research Site, Embourg, Belgium
  - Research Site, Genk, Belgium
  - Research Site, Genly, Belgium
  - Research Site, Gozée, Belgium
  - Research Site, Grivegnée, Belgium
  - Research Site, Halen, Belgium
  - Research Site, Hasselt, Belgium
  - Research Site, Heurne, Belgium
  - Research Site, Heusden, Belgium
  - Research Site, Hove, Belgium
  - Research Site, Kessel-Lo, Belgium
  - Research Site, Kraainem, Belgium
  - Research Site, Landen, Belgium
  - Research Site, Leopoldsburg, Belgium
  - Research Site, Leuven, Belgium
  - Research Site, Libin, Belgium
  - Research Site, Linkebeek, Belgium
  - Research Site, Lommel, Belgium
  - Research Site, Marchienne-au-Pont, Belgium
  - Research Site, Marchovelette, Belgium
  - Research Site, Mechelen-aan-de-Maas, Belgium
  - Research Site, Melsbroek, Belgium
  - Research Site, Mont-sur-Marchienne, Belgium
  - Research Site, Moorsel, Belgium
  - Research Site, Mouscron, Belgium
  - Research Site, Natoye, Belgium
  - Research Site, Oostham, Belgium
  - Research Site, Opgrimbie (maasmechelen), Belgium
  - Research Site, Paal, Belgium
  - Research Site, Puurs, Belgium
  - Research Site, Ronquières, Belgium
  - Research Site, Ronse, Belgium
  - Research Site, Rumst, Belgium
  - Research Site, Saint-Médard, Belgium
  - Research Site, Sint-Gillis-Waas, Belgium
  - Research Site, Steenokkerzeel, Belgium
  - Research Site, Tavier, Belgium
  - Research Site, Tessenderlo, Belgium
  - Research Site, Thuin, Belgium
  - Research Site, Tremelo, Belgium
  - Research Site, Trois-Ponts, Belgium
  - Research Site, Turnhout, Belgium
  - Research Site, Vilvoorde, Belgium
  - Research Site, Waremme, Belgium
  - Research Site, Weerde, Belgium
  - Research Site, Wezembeek-Oppem, Belgium
  - Research Site, Zoersel, Belgium
  - Research Site, Ans
  - Research Site, Brussels
  - Research Site, De Pinte
  - Research Site, Ekeren
  - Research Site, Evergem
  - Research Site, Lauwe
  - Research Site, Massemen
  - Research Site, Moerkerke
  - Research Site, Oudenaarde
  - Research Site, Schoonaarde
  - Research Site, Schuiferskapelle
  - Research Site, Tielt
- Brazil (14):
  - Research Site, Maceió, Alagoas
  - Research Site, Fortaleza, Ceará
  - Research Site, Salvador, Estado de Bahia
  - Research Site, Goiagoianiania, Goiás
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Botucatu, São Paulo
  - Research Site, S.j.rio Preto, São Paulo
  - Research Site, Santos, São Paulo
  - Research Site, São José do Rio Preto, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Campinas
- Bulgaria (8):
  - Research Site, Dimitrovgrad
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Canada (85):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Chilliwack, British Columbia
  - Research Site, Coquitlam, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Langley, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Penticton, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Portage la Prairie, Manitoba
  - Research Site, Winnipeg, Manitoba
  - Research Site, Grand Bay-Westfield, New Brunswick
  - Research Site, Moncton, New Brunswick
  - Research Site, Nackawic, New Brunswick
  - Research Site, Saint John, New Brunswick
  - Research Site, Woodstock, New Brunswick
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Carbonear, Newfoundland and Labrador
  - Research Site, Conception Bay South, Newfoundland and Labrador
  - Research Site, Holyrood, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Amherst, Nova Scotia
  - Research Site, Antigonish, Nova Scotia
  - Research Site, Digby, Nova Scotia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Windsor, Nova Scotia
  - Research Site, Bolton, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Corunna, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Exeter, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Ingersoll, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Niagara Falls, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, North York, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Perth, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Renfrew, Ontario
  - Research Site, Saint Catherines, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Smith Falls, Ontario
  - Research Site, Stirling, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Tillsonburg, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Charlottetown, Prince Edward Island
  - Research Site, Chicoutimi, Quebec
  - Research Site, Courcelette, Quebec
  - Research Site, Drummonville, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, LaSalle, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Georges, Quebec
  - Research Site, Saint-Marc-des-Carrieres, Quebec
  - Research Site, Sainte-Catherine, Quebec
  - Research Site, Sainte-Julie, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Vanier, Quebec
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- Chile (2):
  - Research Site, Temuco, Región de la Araucanía
  - Research Site, Santiago, Santiago Metropolitan
- Colombia (8):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bogotá, Colombia
  - Research Site, Cartagena, Departamento de Bolívar
  - Research Site, Pereira, Risaralda Department
  - Research Site, Bucaramanga, Santander Department
  - Research Site, Floridablanca, Santander Department
  - Research Site, Cali, Valle del Cauca Department
- Costa Rica (4):
  - Research Site, Desamparados, Provincia de San José
  - Research Site, Escazú, Provincia de San José
  - Research Site, San Pedro, Provincia de San José
  - Research Site, Heredia
- Denmark (5):
  - Research Site, Gentofte Municipality
  - Research Site, Glostrup Municipality
  - Research Site, Herlev
  - Research Site, Hillerød
  - Research Site, Odense C
- El Salvador (2):
  - Research Site, El Salvador, San Salvador Department
  - Research Site, San Salvador
- Estonia (6):
  - Research Site, Saku, Harju
  - Research Site, Pärnu
  - Research Site, Rakvere
  - Research Site, Tallinn
  - Research Site, Tartu
  - Research Site, Viljandi County
- Germany (14):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Chemnitz
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Görlitz
  - Research Site, Hamburg
  - Research Site, Künzing
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Nuremberg
  - Research Site, Ulm
  - Research Site, Witten
- Israel (11):
  - Research Site, Kiryat Hadassah, Jerusalem
  - Research Site, Ashkelon Shore
  - Research Site, Beer Yakov
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Zrifin
- Mexico (6):
  - Research Site, Aguascalientes, Aguascalientes
  - Research Site, Mexico City, D.F
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Culiacán, Sinaloa
- Netherlands (17):
  - Research Site, Alkmaar
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Deventer
  - Research Site, Eindhoven
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Hoorn
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, The Hague
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Velp
  - Research Site, Zoetermeer
- Norway (32):
  - Research Site, Bekkestua
  - Research Site, Bergen
  - Research Site, Bøverbru
  - Research Site, Elverum
  - Research Site, Flatåsen
  - Research Site, Fredrikstad
  - Research Site, Halden
  - Research Site, Heimdal
  - Research Site, Kristiansand
  - Research Site, Laksevåg
  - Research Site, Lena
  - Research Site, Lierskogen
  - Research Site, Lysaker
  - Research Site, Løvenstad
  - Research Site, Moelv
  - Research Site, Moss
  - Research Site, Oslo
  - Research Site, Paradis
  - Research Site, Randaberg
  - Research Site, Rådal
  - Research Site, Skedsmokorset
  - Research Site, Ski
  - Research Site, Skiptvet
  - Research Site, Snaroya
  - Research Site, Sogndal
  - Research Site, Spikkestad
  - Research Site, Stavanger
  - Research Site, Strømmen
  - Research Site, Svelvik
  - Research Site, Trollåsen
  - Research Site, Trondheim
  - Research Site, Østerås
- Research Site, Panama City, Provincia de Panamá, Panama
- Poland (42):
  - Research Site, Aleksandrów Łódzki
  - Research Site, Bydgoszcz
  - Research Site, Bytom
  - Research Site, Chodzież
  - Research Site, Chorzów
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Jelcz Laskowice
  - Research Site, Karpacz
  - Research Site, Katowice
  - Research Site, Koluszki
  - Research Site, Krakow
  - Research Site, Linia
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Nowogard
  - Research Site, Olsztyn
  - Research Site, Opalenica
  - Research Site, Opole
  - Research Site, Ostrów Wielkopolski
  - Research Site, Oława
  - Research Site, Piekary Śląskie
  - Research Site, Poznan
  - Research Site, Puławy
  - Research Site, Radom
  - Research Site, Radziejów
  - Research Site, Rybnik
  - Research Site, Sieradz
  - Research Site, Skierniewice
  - Research Site, Sobótka
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Słupca
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Trzcianka
  - Research Site, Turek
  - Research Site, Warsaw
  - Research Site, Wąbrzeźno
  - Research Site, Wejherowo
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Puerto Rico (6):
  - Research Site, Aguas Buenas
  - Research Site, Caguas
  - Research Site, Cidra
  - Research Site, Levittown-toa Baja
  - Research Site, Ponce
  - Research Site, San Juan
- Romania (4):
  - Research Site, Cluj-Napoca, Cluj
  - Research Site, Timișoara, Timiș County
  - Research Site, Brasov
  - Research Site, Bucharest
- Russia (12):
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tolyatti
  - Research Site, Tomsk
  - Research Site, Tyumen
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Africa (19):
  - Research Site, Claremont, Cape Province
  - Research Site, Athlone, Cape Town
  - Research Site, Florida Park, Gauteng
  - Research Site, Lenasia, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Witbank, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, eMkhomazi, KwaZulu-Natal
  - Research Site, Morningside Manor, Morningside
  - Research Site, Korsten, Port Elizabeth
  - Research Site, Hillcrest, Pretoria
  - Research Site, Halfway House, South Africa
  - Research Site, Johannesburg, South Africa
  - Research Site, Worcester, South Africa
  - Research Site, Benoni
  - Research Site, Lakeview, Retreat
  - Research Site, Rustenburg
  - Research Site, Somerset West
  - Research Site, Vanderbijlpark
- Research Site, Olten, Schweiz, Switzerland
- United Kingdom (29):
  - Research Site, Reading, Berkshire
  - Research Site, Annan, Dumfries and Galloway
  - Research Site, Blantyre, Lanarkshire
  - Research Site, Hamilton, Lanarkshire
  - Research Site, Strathaven, Lanarkshire
  - Research Site, Wishaw, Lanarkshire
  - Research Site, Paisley, Renfrewshire
  - Research Site, Airdrie, Scotland
  - Research Site, Glasgow, Scotland
  - Research Site, Barrhead
  - Research Site, Bellshill
  - Research Site, Birmingham
  - Research Site, Cambuslang
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Cumbernauld
  - Research Site, Gourock
  - Research Site, Greenock
  - Research Site, Helensburgh
  - Research Site, Kirkintilloch
  - Research Site, Liverpool
  - Research Site, Lockerbie
  - Research Site, Manchester
  - Research Site, New Stevenson
  - Research Site, Renfrew
  - Research Site, Stranraer
  - Research Site, Strathblane
  - Research Site, Thornhill
  - Research Site, Wolverhampton
- Research Site, Montevideo, Uruguay
- Venezuela (12):
  - Research Site, Maracay, Municipio Girardot, Aragua
  - Research Site, Barinas, Barinas
  - Research Site, Ciudad Bolívar, Bolívar
  - Research Site, Puerto Ordaz and San Felix, Bolívar
  - Research Site, Valencia, Carabobo
  - Research Site, Barquisimeto, Lara
  - Research Site, Latrinidad Caracas, Municipio Baruta
  - Research Site, Mérida, Mérida
  - Research Site, Porlamar, Nueva Esparta
  - Research Site, Punto Fijo, Estado Falcon, Venezuela
  - Research Site, Maracaibo, Zulia
  - Research Site, Caracas

REFERENCES:
- [Derived] Hoshi RA, Alotaibi M, Liu Y, Watrous JD, Ridker PM, Glynn RJ, Serhan CN, Luttmann-Gibson H, Moorthy MV, Jain M, Demler OV, Mora S. One-Year Effects of High-Intensity Statin on Bioactive Lipids: Findings From the JUPITER Trial. Arterioscler Thromb Vasc Biol. 2024 Jul;44(7):e196-e206. doi: 10.1161/ATVBAHA.124.321058. Epub 2024 Jun 6. PMID 38841856
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Ajala ON, Demler OV, Liu Y, Farukhi Z, Adelman SJ, Collins HL, Ridker PM, Rader DJ, Glynn RJ, Mora S. Anti-Inflammatory HDL Function, Incident Cardiovascular Events, and Mortality: A Secondary Analysis of the JUPITER Randomized Clinical Trial. J Am Heart Assoc. 2020 Sep;9(17):e016507. doi: 10.1161/JAHA.119.016507. Epub 2020 Aug 15. PMID 32799709
- [Derived] Akinkuolie AO, Lawler PR, Chu AY, Caulfield M, Mu J, Ding B, Nyberg F, Glynn RJ, Ridker PM, Hurt-Camejo E, Chasman DI, Mora S. Group IIA Secretory Phospholipase A2, Vascular Inflammation, and Incident Cardiovascular Disease. Arterioscler Thromb Vasc Biol. 2019 Jun;39(6):1182-1190. doi: 10.1161/ATVBAHA.118.311894. PMID 31070471
- [Derived] Dagenais GR, Jung H, Lonn E, Bogaty PM, Dehghan M, Held C, Avezum A, Jansky P, Keltai M, Leiter LA, Lopez-Jaramillo P, Toff WD, Bosch J, Yusuf S. Effects of Lipid-Lowering and Antihypertensive Treatments in Addition to Healthy Lifestyles in Primary Prevention: An Analysis of the HOPE-3 Trial. J Am Heart Assoc. 2018 Jul 22;7(15):e008918. doi: 10.1161/JAHA.118.008918. PMID 30033433
- [Derived] Khera AV, Demler OV, Adelman SJ, Collins HL, Glynn RJ, Ridker PM, Rader DJ, Mora S. Cholesterol Efflux Capacity, High-Density Lipoprotein Particle Number, and Incident Cardiovascular Events: An Analysis From the JUPITER Trial (Justification for the Use of Statins in Prevention: An Intervention Trial Evaluating Rosuvastatin). Circulation. 2017 Jun 20;135(25):2494-2504. doi: 10.1161/CIRCULATIONAHA.116.025678. Epub 2017 Apr 27. PMID 28450350
- [Derived] Akinkuolie AO, Glynn RJ, Padmanabhan L, Ridker PM, Mora S. Circulating N-Linked Glycoprotein Side-Chain Biomarker, Rosuvastatin Therapy, and Incident Cardiovascular Disease: An Analysis From the JUPITER Trial. J Am Heart Assoc. 2016 Jul 13;5(7):e003822. doi: 10.1161/JAHA.116.003822. PMID 27413042
- [Derived] Dugani SB, Akinkuolie AO, Paynter N, Glynn RJ, Ridker PM, Mora S. Association of Lipoproteins, Insulin Resistance, and Rosuvastatin With Incident Type 2 Diabetes Mellitus : Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2016 May 1;1(2):136-45. doi: 10.1001/jamacardio.2016.0096. PMID 27347563
- [Derived] Lawler PR, Akinkuolie AO, Chandler PD, Moorthy MV, Vandenburgh MJ, Schaumberg DA, Lee IM, Glynn RJ, Ridker PM, Buring JE, Mora S. Circulating N-Linked Glycoprotein Acetyls and Longitudinal Mortality Risk. Circ Res. 2016 Apr 1;118(7):1106-15. doi: 10.1161/CIRCRESAHA.115.308078. Epub 2016 Mar 7. PMID 26951635
- [Derived] Mora S, Caulfield MP, Wohlgemuth J, Chen Z, Superko HR, Rowland CM, Glynn RJ, Ridker PM, Krauss RM. Atherogenic Lipoprotein Subfractions Determined by Ion Mobility and First Cardiovascular Events After Random Allocation to High-Intensity Statin or Placebo: The Justification for the Use of Statins in Prevention: An Intervention Trial Evaluating Rosuvastatin (JUPITER) Trial. Circulation. 2015 Dec 8;132(23):2220-9. doi: 10.1161/CIRCULATIONAHA.115.016857. Epub 2015 Sep 25. PMID 26408274
- [Derived] Chu AY, Giulianini F, Barratt BJ, Ding B, Nyberg F, Mora S, Ridker PM, Chasman DI. Differential Genetic Effects on Statin-Induced Changes Across Low-Density Lipoprotein-Related Measures. Circ Cardiovasc Genet. 2015 Oct;8(5):688-95. doi: 10.1161/CIRCGENETICS.114.000962. Epub 2015 Aug 13. PMID 26273092
- [Derived] Everett BM, Zeller T, Glynn RJ, Ridker PM, Blankenberg S. High-sensitivity cardiac troponin I and B-type natriuretic Peptide as predictors of vascular events in primary prevention: impact of statin therapy. Circulation. 2015 May 26;131(21):1851-60. doi: 10.1161/CIRCULATIONAHA.114.014522. Epub 2015 Mar 30. PMID 25825410
- [Derived] Everett BM, Mora S, Glynn RJ, MacFadyen J, Ridker PM. Safety profile of subjects treated to very low low-density lipoprotein cholesterol levels (<30 mg/dl) with rosuvastatin 20 mg daily (from JUPITER). Am J Cardiol. 2014 Dec 1;114(11):1682-9. doi: 10.1016/j.amjcard.2014.08.041. Epub 2014 Sep 16. PMID 25439449
- [Derived] Pena JM, Aspberg S, MacFadyen J, Glynn RJ, Solomon DH, Ridker PM. Statin therapy and risk of fracture: results from the JUPITER randomized clinical trial. JAMA Intern Med. 2015 Feb;175(2):171-7. doi: 10.1001/jamainternmed.2014.6388. PMID 25437881
- [Derived] Khera AV, Everett BM, Caulfield MP, Hantash FM, Wohlgemuth J, Ridker PM, Mora S. Lipoprotein(a) concentrations, rosuvastatin therapy, and residual vascular risk: an analysis from the JUPITER Trial (Justification for the Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin). Circulation. 2014 Feb 11;129(6):635-42. doi: 10.1161/CIRCULATIONAHA.113.004406. Epub 2013 Nov 17. PMID 24243886
- [Derived] Mora S, Glynn RJ, Ridker PM. High-density lipoprotein cholesterol, size, particle number, and residual vascular risk after potent statin therapy. Circulation. 2013 Sep 10;128(11):1189-97. doi: 10.1161/CIRCULATIONAHA.113.002671. Epub 2013 Sep 3. PMID 24002795
- [Derived] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Derived] Mora S, Glynn RJ, Boekholdt SM, Nordestgaard BG, Kastelein JJ, Ridker PM. On-treatment non-high-density lipoprotein cholesterol, apolipoprotein B, triglycerides, and lipid ratios in relation to residual vascular risk after treatment with potent statin therapy: JUPITER (justification for the use of statins in prevention: an intervention trial evaluating rosuvastatin). J Am Coll Cardiol. 2012 Apr 24;59(17):1521-8. doi: 10.1016/j.jacc.2011.12.035. PMID 22516441
- [Derived] Stein EA, Vidt DG, Shepherd J, Cain VA, Anzalone D, Cressman MD. Renal safety of intensive cholesterol-lowering treatment with rosuvastatin: a retrospective analysis of renal adverse events among 40,600 participants in the rosuvastatin clinical development program. Atherosclerosis. 2012 Apr;221(2):471-7. doi: 10.1016/j.atherosclerosis.2011.12.011. Epub 2012 Jan 3. PMID 22304793
- [Derived] Dorresteijn JA, Visseren FL, Ridker PM, Wassink AM, Paynter NP, Steyerberg EW, van der Graaf Y, Cook NR. Estimating treatment effects for individual patients based on the results of randomised clinical trials. BMJ. 2011 Oct 3;343:d5888. doi: 10.1136/bmj.d5888. PMID 21968126
- [Derived] Albert MA, Glynn RJ, Fonseca FA, Lorenzatti AJ, Ferdinand KC, MacFadyen JG, Ridker PM. Race, ethnicity, and the efficacy of rosuvastatin in primary prevention: the Justification for the Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER) trial. Am Heart J. 2011 Jul;162(1):106-14.e2. doi: 10.1016/j.ahj.2011.03.032. Epub 2011 Jun 12. PMID 21742096
- [Derived] Ridker PM, MacFadyen JG, Glynn RJ, Chasman DI. Kinesin-like protein 6 (KIF6) polymorphism and the efficacy of rosuvastatin in primary prevention. Circ Cardiovasc Genet. 2011 Jun;4(3):312-7. doi: 10.1161/CIRCGENETICS.110.959353. Epub 2011 Apr 14. PMID 21493817
- [Derived] Koenig W, Ridker PM. Rosuvastatin for primary prevention in patients with European systematic coronary risk evaluation risk >/= 5% or Framingham risk >20%: post hoc analyses of the JUPITER trial requested by European health authorities. Eur Heart J. 2011 Jan;32(1):75-83. doi: 10.1093/eurheartj/ehq370. Epub 2010 Oct 22. PMID 20971747
- [Derived] Ridker PM, Macfadyen JG, Nordestgaard BG, Koenig W, Kastelein JJ, Genest J, Glynn RJ. Rosuvastatin for primary prevention among individuals with elevated high-sensitivity c-reactive protein and 5% to 10% and 10% to 20% 10-year risk. Implications of the Justification for Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER) trial for "intermediate risk". Circ Cardiovasc Qual Outcomes. 2010 Sep;3(5):447-52. doi: 10.1161/CIRCOUTCOMES.110.938118. Epub 2010 Aug 24. PMID 20736443
- [Derived] Ridker PM, Genest J, Boekholdt SM, Libby P, Gotto AM, Nordestgaard BG, Mora S, MacFadyen JG, Glynn RJ, Kastelein JJ; JUPITER Trial Study Group. HDL cholesterol and residual risk of first cardiovascular events after treatment with potent statin therapy: an analysis from the JUPITER trial. Lancet. 2010 Jul 31;376(9738):333-9. doi: 10.1016/S0140-6736(10)60713-1. Epub 2010 Jul 23. PMID 20655105
- [Derived] Ridker PM, MacFadyen J, Cressman M, Glynn RJ. Efficacy of rosuvastatin among men and women with moderate chronic kidney disease and elevated high-sensitivity C-reactive protein: a secondary analysis from the JUPITER (Justification for the Use of Statins in Prevention-an Intervention Trial Evaluating Rosuvastatin) trial. J Am Coll Cardiol. 2010 Mar 23;55(12):1266-1273. doi: 10.1016/j.jacc.2010.01.020. Epub 2010 Mar 4. PMID 20206456
- [Derived] Mora S, Glynn RJ, Hsia J, MacFadyen JG, Genest J, Ridker PM. Statins for the primary prevention of cardiovascular events in women with elevated high-sensitivity C-reactive protein or dyslipidemia: results from the Justification for the Use of Statins in Prevention: An Intervention Trial Evaluating Rosuvastatin (JUPITER) and meta-analysis of women from primary prevention trials. Circulation. 2010 Mar 9;121(9):1069-77. doi: 10.1161/CIRCULATIONAHA.109.906479. Epub 2010 Feb 22. PMID 20176986
- [Derived] Ridker PM, MacFadyen JG, Fonseca FA, Genest J, Gotto AM, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Number needed to treat with rosuvastatin to prevent first cardiovascular events and death among men and women with low low-density lipoprotein cholesterol and elevated high-sensitivity C-reactive protein: justification for the use of statins in prevention: an intervention trial evaluating rosuvastatin (JUPITER). Circ Cardiovasc Qual Outcomes. 2009 Nov;2(6):616-23. doi: 10.1161/CIRCOUTCOMES.109.848473. Epub 2009 Sep 22. PMID 20031900
- [Derived] Everett BM, Glynn RJ, MacFadyen JG, Ridker PM. Rosuvastatin in the prevention of stroke among men and women with elevated levels of C-reactive protein: justification for the Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER). Circulation. 2010 Jan 5;121(1):143-50. doi: 10.1161/CIRCULATIONAHA.109.874834. Epub 2009 Dec 21. PMID 20026779
- [Derived] Glynn RJ, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Ridker PM. A randomized trial of rosuvastatin in the prevention of venous thromboembolism. N Engl J Med. 2009 Apr 30;360(18):1851-61. doi: 10.1056/NEJMoa0900241. Epub 2009 Mar 29. PMID 19329822
- [Derived] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, Macfadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Trial Study Group. Reduction in C-reactive protein and LDL cholesterol and cardiovascular event rates after initiation of rosuvastatin: a prospective study of the JUPITER trial. Lancet. 2009 Apr 4;373(9670):1175-82. doi: 10.1016/S0140-6736(09)60447-5. Epub 2009 Mar 28. PMID 19329177
- [Derived] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=317&filename=CSR-D3560L00030.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 05 February 2003. The last subject completed on 20 August 2008. Study subjects were randomized at 1348 centers in 26 countries. Enrolled subjects participated in an initial 4-week, run-in phase and received placebo therapy.
Pre-assignment Details: If found eligible for the main study on the basis of appropriate levels of baseline Low Density Lipoprotein (LDL), High-sensitivity C-Reactive Protein (hsCRP), and run-in phase compliance (>80% of pills taken), subjects were randomized to either rosuvastatin 20 mg or placebo once daily
Period: Overall Study
Arm/Group | Rosuvastatin | Placebo
Started | 8901 | 8901
Randomized and Treated (Safety Pop) | 8869 | 8864
Completed | 8208 | 8186
Not Completed | 693 | 715
Not completed — Adverse Event | 100 | 99
Not completed — Withdrawal by Subject | 458 | 489
Not completed — Lost to Follow-up | 28 | 22
Not completed — Protocol Violation | 4 | 4
Not completed — Physician Decision | 13 | 17
Not completed — No information chacked on CaseReportForm | 90 | 84

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Placebo | Total
Number analyzed (Participants) | 8901 | 8901 | 17802
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (7.64) | 66.1 (7.8) | 66.1 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3426 | 3375 | 6801
  Male | 5475 | 5526 | 11001

OUTCOME MEASURES:

1. Primary Outcome: Time to Major Cardiac Event (Cardiovascular Death, Stroke, Myocardial Infarction, Hospitalization Due to Unstable Angina or Arterial Revascularization)
Description: Days from randomization to the first of CV death, stroke, MI, hospitalization for unstable angina or arterial revascularization. If no event, censoring occurs at earliest of termination date or efficacy cut-off date of 30 Mar 2008. Events were adjudicated by an endpoint committee. Kaplan-Meier estimate of the mean
Time Frame: up to 5 years
Population: Intention to treat population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 8901 | 8901
Days | 1646.4 (2.76) | 1578.3 (3.49)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.56, 95% CI [0.46 to 0.69] — The hazard ratio shows (Rosuvastatin hazard/Placebo hazard)

2. Secondary Outcome: Time to Death Due to Any Cause
Description: Days from randomization to death. If no death then censoring occurs at earliest of termination date or efficacy cutoff date of 30 Mar 2008. Kaplan-Meier estimate of the mean
Time Frame: up to 5 years
Population: Intention to treat population
Measure: Mean (Standard Error); unit: days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 8901 | 8901
days | 1543.3 (2.48) | 1619.1 (3.10)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p < 0.021, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI [0.67 to 0.97] — The hazard ratio shows (Rosuvastatin hazard/Placebo hazard)

3. Secondary Outcome: Time to Non-cardiovascular Death
Description: Days from randomization to death from a non-cardiovascular cause. If no event, then censoring occurs at earliest of termination date or efficacy cutoff date of 30 Mar 2008. Events were adjudicated by an endpoint committee. Kaplan-Meier estimate of the mean
Time Frame: up to 5 years
Population: Intention to treat population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 8901 | 8901
Days | 1558.5 (1.90) | 1640.5 (2.44)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p < 0.172, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI [0.65 to 1.08] — The hazard ratio shows (Rosuvastatin hazard/Placebo hazard)

4. Secondary Outcome: Time to Development of Diabetes Mellitus
Description: Days from randomization until development of diabetes. If no diabetes was developed censoring occurred at termination date. Kaplan-Meier estimate of the mean
Time Frame: up to 5 years
Population: Intention to treat population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 8901 | 8901
Days | 1687.0 (3.92) | 1517.0 (2.46)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p < 0.015, Regression, Cox; Hazard Ratio (HR) = 1.27, 95% CI [1.05 to 1.53] — The hazard ratio shows (Rosuvastatin hazard/Placebo hazard)

5. Secondary Outcome: Time to Venous Thromboembolic Event
Description: Time from randomization to the first venous thromboembolic event. Kaplan-Meier estimate of the mean
Time Frame: up to 5 years
Population: Intention to treat population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 8901 | 8901
Days | 1147.4 (0.54) | 1377.2 (1.05)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p = 0.018, Regression, Cox; Hazard Ratio (HR) = 0.57, 95% CI [0.35 to 0.91] — The hazard ratio shows (Rosuvastatin hazard/Placebo hazard)

6. Secondary Outcome: Time to Bone Fracture
Description: Days from randomization until bone fracture. If no event, then censoring occurs at earliest of termination date or efficacy cutoff date of 30 Mar 2008. Kaplan-Meier estimate of the mean
Time Frame: Up to 5 years
Population: Intention to treat population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 8901 | 8901
Days | 1662.7 (3.35) | 1546.9 (2.78)
Statistical Analysis 1: Comparison: Rosuvastatin vs Placebo; Test type: Superiority or Other; p = 0.548, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI [0.88 to 1.28] — The hazard ratio shows (Rosuvastatin hazard/Placebo hazard)

ADVERSE EVENTS:
Arm/Group | PLACEBO | ROSUVASTATIN 20 MG
Serious Adverse Events (participants affected / at risk) | 1216/8864 | 1205/8869
Other Adverse Events (participants affected / at risk) | 3170/8864 | 3228/8869
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=8864) | ROSUVASTATIN 20 MG (N=8869)
Anaemia (Blood and lymphatic system disorders) | 11 (11) | 15 (15)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pernicious anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
AV dissociation (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 10 (10) | 10 (10)
Angina unstable (Cardiac disorders) | 6 (6) | 3 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 65 (65) | 56 (56)
Atrial flutter (Cardiac disorders) | 9 (9) | 5 (5)
Atrial tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 5 (5)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 6 (6) | 10 (10)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 5 (5) | 6 (6)
Cardiac failure congestive (Cardiac disorders) | 19 (19) | 16 (16)
Cardiac valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 3 (3) | 2 (2)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 3 (3)
Myocardial infarction (Cardiac disorders) | 7 (7) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 6 (6) | 5 (5)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular flutter (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Congenital intestinal malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Duchenne muscular dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Lymphangioma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Auricular swelling (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vestibular neuronitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 4 (4)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Pituitary cyst (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 2 (2)
Thyroid mass (Endocrine disorders) | 2 (2) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 8 (8) | 3 (3)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Ectropion (Eye disorders) | 0 (0) | 1 (1)
Endophthalmitis (Eye disorders) | 0 (0) | 2 (2)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Lacrimal disorder (Eye disorders) | 0 (0) | 1 (1)
Lenticular opacities (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 3 (3) | 3 (3)
Retinal tear (Eye disorders) | 2 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 9 (9)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (4)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 2 (2) | 0 (0)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colonic polyp (Gastrointestinal disorders) | 3 (3) | 4 (4)
Colonic stenosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 5 (5)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 2 (2)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (13) | 20 (20)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 3 (3)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 4 (4)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 15 (15) | 17 (17)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 11 (11)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 6 (6) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 6 (6) | 9 (9)
Pancreatolithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland cyst (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (7) | 5 (5)
Spigelian hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 5 (5) | 8 (8)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Adhesion (General disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Calcinosis (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 7 (7) | 9 (9)
Death (General disorders) | 34 (34) | 30 (30)
Deformity (General disorders) | 1 (1) | 0 (0)
Dysplasia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 2 (2) | 2 (2)
Hernia obstructive (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 22 (22) | 29 (29)
Oedema peripheral (General disorders) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 4 (4)
Sudden death (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Ulcer (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 5 (5) | 4 (4)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 9 (9) | 10 (10)
Cholecystitis acute (Hepatobiliary disorders) | 5 (5) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 4 (4) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 23 (23) | 22 (22)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cyst ruptured (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 4 (4)
Sarcoidosis (Immune system disorders) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Abscess rupture (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 7 (7) | 5 (5)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 3 (3) | 1 (1)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 5 (5) | 7 (7)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 3 (3) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 20 (20) | 13 (13)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Corneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 16 (16) | 13 (13)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 11 (11) | 8 (8)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Incision site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 9 (9) | 4 (4)
Lung abscess (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Meningococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Parotid abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 57 (57) | 56 (56)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 2 (2)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 11 (11)
Septic shock (Infections and infestations) | 2 (2) | 4 (4)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Subacute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 3 (3)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 15 (15)
Urosepsis (Infections and infestations) | 4 (4) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 2 (2)
Viral pericarditis (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (4) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 9 (9) | 14 (14)
Back injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Caustic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Crush injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 6 (6) | 8 (8)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 14 (14) | 15 (15)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Retinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
Road traffic accident (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Anticonvulsant drug level increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 13 (13) | 14 (14)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Lipomatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 53 (53) | 48 (48)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Bunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 (12) | 9 (9)
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 15 (15) | 17 (17)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 11 (11)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 5 (5)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (22) | 20 (20)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (20) | 16 (16)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5)
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 10 (10)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 7 (7)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 38 (38) | 34 (34)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pseudomyxoma peritonei (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Ureteric cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 (2) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anticholinergic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 9 (9)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3)
Drop attacks (Nervous system disorders) | 1 (1) | 0 (0)
Drug withdrawal convulsions (Nervous system disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 3 (3)
Facial neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 1 (1) | 2 (2)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hemicephalalgia (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 2 (2) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myxoedema coma (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 2 (2) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 5 (5)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 2 (2)
Senile dementia (Nervous system disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 15 (15) | 11 (11)
Transient ischaemic attack (Nervous system disorders) | 10 (10) | 9 (9)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 7 (7)
Delirium (Psychiatric disorders) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 7 (7)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 5 (5) | 0 (0)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (6) | 11 (11)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 12 (12) | 7 (7)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 4 (4) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 7 (7) | 6 (6)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 6 (6)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 5 (5) | 7 (7)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 2 (2)
Vesical fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 17 (17) | 12 (12)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 5 (5) | 3 (3)
Rectocele (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cervical erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 4 (4) | 7 (7)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 25 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Eosinophilic pneumonia chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 11 (11)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (12)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Facial hemiatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Pancreatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 5 (5) | 3 (3)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 4 (4)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 13 (13) | 7 (7)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 7 (7) | 9 (9)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 2 (2)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 2 (2) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 2 (2) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 2 (2)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=8864) | ROSUVASTATIN 20 MG (N=8869)
Bronchitis (Infections and infestations) | 571 (571) | 596 (596)
Nasopharyngitis (Infections and infestations) | 607 (607) | 632 (632)
Upper respiratory tract infection (Infections and infestations) | 637 (637) | 580 (580)
Urinary tract infection (Infections and infestations) | 686 (686) | 699 (699)
Back pain (Musculoskeletal and connective tissue disorders) | 576 (576) | 631 (631)
Myalgia (Musculoskeletal and connective tissue disorders) | 559 (559) | 653 (653)
Hypertension (Vascular disorders) | 628 (628) | 557 (557)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No